CLINICAL TRIAL: NCT06037343
Title: Deep Learning Image Reconstruction for Abdominal CT of Hepatocellular Carcinoma Compared With 3-TESLA MRI
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Valérie LAURENT, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI111
Record Dates: First submitted 2023-08-31; First posted 2023-09-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; DLIR CT; ASIR reconstruction
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
New algorithms for processing CT acquisitions, based on artificial intelligence, have been reported to improve acquisition quality. Thats' why it's possible to imagine that new scan post-processing algorithms enable better detection and characterization of hepatocellular carcinoma lesions than with standard reconstructions. DLIR reconstructions could even match with MRI detection.

The aim of the study is to compare the detection and characterization of hepatic lesions according to the LI-RADS classification in CT with DLIR artificial intelligence reconstruction, compared with ASIR-V reconstruction and the gold standard of MRI.

ELIGIBILITY:
Inclusion Criteria:

* undergoing CT and MRI scans in the same week, with protocols dedicated to the detection of HCC lesions

Exclusion Criteria:

* imaging with radiological artefact

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adults undergoing a CT and a MRI for detection or following of an HCC during the same week
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Lesion size in mm | Through study completion, an average of 1 year
Hypervascular appearance of lesion | Through study completion an average of 1 year
  Qualitative measurement: presence or absence of hypervascular lesion
Hypervascular capsule | Through study completion an average of 1 year
  Qualitative measurement : presence or absence of hypervascular capsule

SECONDARY OUTCOMES:
Infiltrative nature Classification of the hepatic lesion by LI-RADS in MRI | Through study completion an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No